CLINICAL TRIAL: NCT06553859
Title: Prospective Observational Study to Evaluate the Effect of Supercritical Carbon Dioxide-Processed Acellular Dermal Matrix (SC Derm® Recon) in Prosthetic Breast Reconstruction
Brief Title: Evaluation of ADM(SC Derm® Recon) in Breast Reconstruction
Acronym: SCderm
Status: Recruiting | Type: Observational
Sponsor: DOF Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-01-001
Record Dates: First submitted 2024-07-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Female
Keywords: Breast Reconstruction using Implants and ADM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: Fifty subjects are to be enrolled prospectively. Breast cancer patients who are willing to undergo breast reconstruction surgery based on inserting breast implants with ADM will be selected as the test group, with "SC Derm"(Acellular Dermal Matrix processed by CO2 supercritical fluid technology.)
  Interventions: Other: No intervention conducts.
- Control Group: Fifty subjects are to be enrolled retrospectively from the medical records of breast cancer patients who have undergone breast reconstruction surgery based on inserting breast implants with ADM made by other companies. All breast reconstruction surgeries have operated from 1, June 2021 to 9, November 2021 at Asan medical center at Seoul, South Korea.

INTERVENTIONS:
Other: No intervention conducts. — The type and method of breast reconstruction with sillicon implants and ADM implanting is now the standard treatment of breast cancer in korea. no any specific intervention has occurred during the surgery.
  Groups: Test Group

SUMMARY:
The goal of this observational study is to examine any clinical differences in the outcomes of breast reconstruction surgeries using Acellular Dermal Matrix (ADM) processed by CO2 supercritical fluid technology compared to other ADM products that have been washed with detergents. The study will also assess safety outcomes.

DETAILED DESCRIPTION:
The total number of study subjects is 100, with 50 people recruited prospectively into the test group and 50 people retrospectively into the control group.

The test group will consist of 50 patients aged 20 to 80 who have undergone total mastectomy for breast cancer and are scheduled to undergo immediate breast reconstruction using implants. These subjects will receive SC Derm (ADM processed by DOF Inc.) during the implant-based breast reconstruction surgery.

The control group will consist of 50 patients who will be retrospectively and consecutively selected from medical records of patients who underwent implant breast reconstruction using ADM from other companies between June 1, 2021, and November 9, 2021.

Patients who fall into the following categories cannot participate in this clinical study because they meet the exclusion criteria:

1. Patients who have received an organ transplant and are taking any immunosuppressants.
2. Patients whose mental condition may affect the progress of the clinical study due to alcohol or drug abuse.
3. Individuals who are unable to complete the survey conducted in this clinical study.
4. Patients who participated in other clinical trials within the previous 120 days at the time of screening.
5. Patients for whom the investigator determines participation in the study is not appropriate.

Among breast cancer patients who decide to undergo implant-based breast reconstruction after total mastectomy at our hospital, the investigator will fully explain the study to these patients during outpatient visits and recruit those who voluntarily express their willingness to participate.

Before any screening or enrollment, all subjects must confirm their willingness to participate by signing the informed consent form.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 to 80 who undergo immediate breast reconstruction using implants after taking total mastectomy

Exclusion Criteria:

Patients who fall into the five categories below cannot participate in this clinical study because they meet the exclusion criteria for research subjects.

1. Patients who have received an organ transplant and are taking any immunosuppressant.
2. Patients whose mental condition may affect the progress of clinical study due to alcohol or drug abuse.
3. People who are unable to complete the survey conducted in this clinical study.
4. Patients who participated in other clinical trials within the previous 120 days at the time of screening.
5. If the investigator determine for a patient not to participate this clinical study since participation of the study is not appropriate.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is scheduled to include 50 prospective and 50 retrospective subjects. The retrospective recruitment period for subjects is from June 1, 2021 to November 9, 2021. Patients who meet the inclusion criteria will be consecutively selected from patients who underwent breast reconstruction with implants. The basis for calculation of retrospective patients was not statistically calculated, but considering that the number of implant breast reconstruction patients at our hospital is 500 per year, when only patients who completed follow-up for more than 1 year were included, approximately 5-10% were enrolled in the study. This was expected and calculated to be possible.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The number of occurrences of pre-determined expected adverse events and complications | From the day of operation of breast reconstruction to 12 months
  The number of occurrences of pre-determined expected adverse reactions and complications will be compared between the experimental group and the control group.

SECONDARY OUTCOMES:
Subjects' self-assessment of satisfaction with physical and psychological well-being using the BREAST-Q survey | From the day of operation of breast reconstruction to 12 months
  Subjects will complete the BREAST-Q survey before and after breast reconstruction surgery, which includes multiple questions on a scale from 1 to 5, where a higher score represents greater satisfaction. For instance, there is a question from the satisfaction with breasts part "In the past week, how satisfied or dissatisfied were you with how you look in the mirror with clothes on?" The answer would be selected the scale from 1 (Very Dissatisfied) to 4 (Very Satisfied). The evaluation will be implemented by comparison of average scores for each question between the experimental group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsup Um, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mazari FAK, Wattoo GM, Kazzazi NH, et al. The comparison of strattice and surgimend in acellular dermal matrix-assisted, implant-based immediate breast reconstruction. Plast Reconstr Surg 2018;141(2):283-293 — https://pubmed.ncbi.nlm.nih.gov/29369979/
- See also: Polotto S, Bergamini ML, Pedrazzi G, et al. One-step prepectoral breast reconstruction with porcine dermal matrix-covered implant: a protective technique improving the outcome in post-mastectomy radiation therapy setting. Gland Surg 2020;9(2):219-228 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7225454/
- See also: Decreased length of postoperative drain use, parental opioids, length of stay and complication rates in patients receiving meshed versus unmeshed acellular dermal matrix in 194 submuscular tissue expander-based breast reconstructions — https://pubmed.ncbi.nlm.nih.gov/32221196/
- See also: Viezel-Mathieu A, Alnaif N, Aljerian A, et al.Acellualr dermal matrix-sparing direct-to-implant prepectoral breast reconstruction: A comparative study including cost analysis. Ann Plast Surg 2020;84(2):139-143 — https://pubmed.ncbi.nlm.nih.gov/31335468/
- See also: Nam SY, Youn D, Kim GH, et al. In vitro characterization of a novel human acellular dermal matrix(BellaCell HD) for breast reconstruction. Bioengineering(Basel) 2020;7(2):39. — https://pubmed.ncbi.nlm.nih.gov/32353944/
- See also: Seo Y, Jung Y, Kim SH. Decellularized heart ECM hydrogel using supercritical carbon dioxide for improved angiogenesis. Acta Biomater. 2018;67:270-281 — https://pubmed.ncbi.nlm.nih.gov/29223704/